CLINICAL TRIAL: NCT02929290
Title: Safety, Efficacy and Pharmacokinetic of BPI-9016M in Patients With c-Met- Dysregulated Advanced NSCLC: A Phase Ib Study,Open-label,Dose-expansion Study
Brief Title: Safety, Efficacy and Pharmacokinetic of BPI-9016M in Patients With c-Met- Dysregulated Advanced NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-CM-I02
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPI-9016M (Experimental): Part I：Four dose cohorts will be evaluated, including 300mg, 450mg, 600mg, 800mg. BPI-9016M Tablet will be administered orally to patients once daily for each dose cohort.
  Part II：400mg BPI-9016M Tablet will be administered orally to patients twice a day.
  Interventions: Drug: BPI-9016M

INTERVENTIONS:
Drug: BPI-9016M — Part I：Four dose cohorts will be evaluated, including 300mg, 450mg, 600mg, 800mg. BPI-9016M Tablet will be administered orally to patients once daily for each dose cohort.
  Part II：400mg BPI-9016M Tablet will be administered orally to patients twice a day.
  Other Names: No other name so far

SUMMARY:
The main objective of this study is to evaluate the safety, tolerability, efficacy and pharmacokinetics of BPI-9016M in patients with c-Met-dysregulated advanced NSCLC. Biomarkers related to the efficacy of BPI-9016M will be investigated.

DETAILED DESCRIPTION:
This study was a multicenter, open, single-arm, Ib-stage expanded clinical study.

Part I：On the basis of Ia-stage dose escalation study, a safe and effective dose of -300 mg, 450 mg, 600 mg and 800 mg was selected to enlarge the enrollment study in patients with c-Met-dysregulated advanced NSCLC, and continuously administered until the disease progressed or could not be tolerated, in order to further evaluate the safety, ttolerability, efficacy and pharmacokinetics of BPI-9016M.

Part II：On the basis of the completed research results of Ia stage and part I, a safe and effective dose of 400 mg twice a day (bid) was selected to conduct an expanded enrollment study in NSCLC patients with MET exon 14 skipping alterations, and continuously administered until the disease progressed or could not be tolerated, in order to further evaluate the safety, ttolerability, efficacy and pharmacokinetics of BPI-9016M.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, locally advanced or metastatic NSCLC patients, who is not suitable for surgery or radiotherapy
* Evaluable or measurable disease per Response Evaluation Criteria in Solid Tumors(RECIST1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy ≥12 weeks
* Must have evidence of positive c-Met protein expression by IHC from either local data or the results of molecular pre-screening evaluations；Must haved evidence of MET exon 14 skipping alterations in blood and/or tissue samples.
* Adequate bone marrow, hepatic, and renal function
* Patients of child bearing potential must agree to take contraception during the study and for 3 months after the last day of treatment
* Signed Informed Consent Form

Exclusion Criteria:

* Prior or current treatment with the type II of c-MET inhibitor or HGF/c-Met antibody therapy
* Confirmed ALK or ROS1 rearrangement
* Prior treatment with targeting agents (Including EGFR tyrosine kinase inhibitors,VEGFR TKIs,the tpye I of MET TKIs, etc.) within 14 days or 5 half-life
* Prior treatment with anticancer agents (Including cytotoxic chemotherapy,radiotherapy, immunotherapy etc.) within 4 weeks
* Brain/meninges metastases unless asymptomatic, stable and not requiring steroids for maintenance
* History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease, radiological documentation of idiopathic pulmonary fibrosis at baseline; uncontrolled pleural effusion/pericardial effusion
* Any evidence of severe or uncontrolled systemic diseases, including CTCAE 2 or higher active infection, unstable angina pectoris, congestive cardiac failure and severe liver/renal or metabolic disease
* Active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV)
* History of organ transplant; had surgery or severe injury within 4 weeks
* Uncontrolled hypertension（Systolic blood pressure≥160mmHg and/or diastolic blood pressure≥100mmHg ）
* Patients unable to swallow orally administered medication, prior surgical procedures affecting absorption.
* Pregnant (positive pregnancy test) or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Participants with Adverse Events | 18 months
Objective Response Rate | 16 weeks
Disease Control Rate | 16 weeks

SECONDARY OUTCOMES:
AUCss | 4 weeks
Css-min | 18 months
Progression-Free Survival | 18 months
Overall Survival | 24 months

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Department of Medical Oncology, Cancer Institute/Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of China Medical University, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu X, Cui X, Wang Z, Liu Y, Luo Y, Zhong W, Zhao H, Yao M, Jiang D, Wang M, Chen M, Zheng X, Ding L, Wang Y, Yuan X, Wu P, Hu B, Han X, Shi Y. Safety, efficacy and pharmacokinetics of BPI-9016M in c-MET overexpression or MET exon 14 skipping mutation patients with locally advanced or metastatic non-small-cell lung cancer: a phase Ib study. BMC Cancer. 2023 Apr 11;23(1):331. doi: 10.1186/s12885-022-10500-y. PMID 37041472